CLINICAL TRIAL: NCT03260075
Title: Effects of the Presence of Ward Cats on Patient Satisfaction and Ward Atmosphere for Patients With Substance Abuse, Depression and Psychosis at UPK Basel
Brief Title: Effects of Ward Cats in Patients With Substance Abuse, Depression and Psychosis at UPK Basel
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00540
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2017-08

CONDITIONS: Satisfaction; Station Atmosphere
MeSH Terms: conditions — Personal Satisfaction | interventions — Catalase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ward cat: Patients and staff at wards that have a cat present
  Interventions: Other: cat
- no ward cat: Patients and staff at wards that have no cat present

INTERVENTIONS:
Other: cat — Cat living at the ward
  Groups: ward cat

SUMMARY:
The aim of this study is to explore the relationship between ward cats and patient satisfaction and stations atmosphere in patients with substance abuse, depression and psychosis. Moreover, we wanted to investigate the patients perception of the ward cats and the relationship between station atmosphere perceived by the employees working wards with and without cat at UKP Basel.

DETAILED DESCRIPTION:
The following tools were used to address these aims:

* Available MüPF data regarding patient satisfaction of 170 inpatients during 2016 was analyzed.
* Available MüPF data regarding patient satisfaction of 151 inpatients during 2017 was analyzed.
* 33 patients were interviewed regarding their perception of the cats
* 30 staff members at the wards filled in questionnaires regarding station atmosphere (EssenCES)

ELIGIBILITY:
Inclusion Criteria:

* Inpatient of the 7 wards at UPK Basel diagnosed with substance abuse, depression and psychosis
* staff working at these wards

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients at UPK Basel diagnosed with substance abuse, depression and psychosis as well as staff members working at these wards.
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction (MüPF) | August - Sept 2017
  Questionnaire MüPF 27

SECONDARY OUTCOMES:
station atmosphere | August - Sept 2017
  Questionnaire EssenCES filled out by staff members
Patient satisfaction (interview) | August - Sept 2017
  Patients ratings of satisfaction is assessed in a semi-structured interview
Patients perception of cats | August - Sept 2017
  Patients perception of cats is assessed in a semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hediger, Dr., Principal Investigator — University of Basel
Locations (1):
- Universitäre Psychiatrische Kliniken Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided